CLINICAL TRIAL: NCT07043166
Title: Epidemiological Survey and Follow-up of Cardiovascular-Kidney-Metabolic Diseases Among Adults in Shanghai
Brief Title: Cardiovascular-Kidney-Metabolic Syndrome in Shanghai Zicitizens
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: STONE
Record Dates: First submitted 2025-06-14; First posted 2025-06-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Syndrome; Diabetes; Obesity and Overweight; Hypertension; Dyslipidemia; Thyroid Diseases; Bone Metabolism Disorder; Chronic Kidney Disease(CKD); Cardiovascular Diseases (CVD); Cardiovascular-kidney-metabolic Syndrome
Keywords: Cardiovascular-Kidney-Metabolic Syndrome; metabolic disorders; screening; risk factor; evaluation; prediction
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity; Overweight; Hypertension; Dyslipidemias; Thyroid Diseases; Bone Diseases, Metabolic; Renal Insufficiency, Chronic; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected at every visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is to conduct follow-up assessments and update the cardiorenal outcomes among the STONE cohort that was established during 2016-2017. The secondary aim is to compare metabolic risk factors, metabolic disturbances, and clinically relevant metabolic outcomes between the follow-up period and the baseline assessment. The exploratory goal is to examine the relationships between changes in risk factors and clinical outcomes in the participants.

The study is planned to begin in May 2025 and will finalize the data collection for the entire population by June 2026. During this time, participants will be categorized based on CKM staging. The follow-up phase will continue until 2035.

DETAILED DESCRIPTION:
Between 2016 and 2017, Shanghai Changzheng Hospital conducted a random stratified sampling in 10 communities in Shanghai among individuals aged 18-65 years who had resided in the community for more than six months. Pregnant women, individuals with fractures, severe mental disorders or dementia, bedridden individuals, and those with hepatitis, tuberculosis, AIDS, other infectious diseases, severe liver or kidney dysfunction, and other serious life-threatening diseases were excluded. The Shanghai Thyroid autOimmuNity: an Epidemiological research (STONE) cohort was established. Trained physicians collected multidimensional baseline health data from more than 4,000 Shanghai community residents through questionnaires, structured interviews, physical examinations, and clinical tests. The data included demographic information (gender, age, education level, marital status, employment status, income level, etc.), lifestyle and psychological status (smoking history, alcohol consumption history, dietary habits, sleep, physical activity, etc.), physical examination indicators (height, weight, waist circumference, blood pressure), comprehensive metabolic indicators (complete blood count, liver and kidney function, thyroid function, glucose metabolism indicators, lipid metabolism indicators, tumor immunity, hormone levels), and ultrasound imaging data (abdominal ultrasound, thyroid ultrasound, carotid ultrasound, bone density).

ELIGIBILITY:
Inclusion Criteria:

1. The 4,094 residents of Shanghai communities who have been enrolled in the STONE cohort.
2. Individuals who completed the baseline questionnaire survey, physical examination, and related clinical tests between 2016 and 2017, with complete data records.
3. Willingness to participate in this follow-up study and provision of informed consent.

Exclusion Criteria:

1. Participants who have moved away from their original community and have been living elsewhere for more than two years.
2. Participants whose contact information has changed or become invalid, resulting in loss of contact (those who remain uncontactable after three attempts to reach out).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 4,094 residents were drawn from 10 communities in Shanghai, with baseline multidimensional data collected."
Sampling Method: Probability Sample
Enrollment: 4094 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2035-05-30 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who developed cardiovascular diseases. | Through study completion, an average of 10 year
  The diagnosis of cardiovascular diseases should be made according to the outcomes of carotid ultrasound and cardiac biomarkers.

SECONDARY OUTCOMES:
Number of Participants Who developed metabolic disorders. | Through study completion, an average of 10 year
  Metabolic disorders include obesity, dyslipidemia, diabetes, fatty liver diseases, hypertension, hyperuricemia, chronic kidney disease, thyroid diseases, and bone metabolism-related disorders.

CONTACTS AND LOCATIONS:
Overall Officials: tuo Li, Prof., Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No